CLINICAL TRIAL: NCT03247010
Title: Characterization of Bone Marrow Suppression and Recovery During Radionuclide Treatment Using Functional Tests of Thrombocytes and Hemostasis
Brief Title: Bone Marrow Suppression and Recovery During Radionuclide Treatment
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marie Øbro Fosbøl, MD, PhD student, Rigshospitalet, Denmark
Other Study IDs: Radium-Trombocyt
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Castration-resistant Prostate Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling — Blood samples are taken before each cycle of Radium 223

SUMMARY:
Radium-223-dichloride is approved therapy for patients with metastatic castration-resistant prostate cancer and bone metastases. More than 20 % of patients treated at Rigshospitalet develop bone marrow suppression as a side effect to Radium therapy The aim of the study is to examine biomarkers of bone marrow suppression and recovery during Radium therapy as well as markers of bone remodeling.

DETAILED DESCRIPTION:
Radium-223-dichloride is approved therapy for patients with metastatic castration-resistant prostate cancer and bone metastases. Therapy is administered intravenously every 4 weeks for up to 6 cycles. More than 20 % of patients treated at Rigshospitalet develop bone marrow suppression as a side effect to Radium therapy, which delays or excludes the patient from further oncological therapy. Especially thrombocytopenia is a frequent side-effect and can be long lasting.

The aim of the study is to examine whether biomarkers of bone marrow recovery (immature platelets, platelet volume, reticulocytes, red cell distribution width) can predict development of hematological toxicity during Radium therapy. Furthermore, to investigate whether these biomarkers can predict recovery from toxicity in patients who develop bone marrow suppression during therapy.

A secondary aim of the study is to evaluate whether dynamics in biomarkers of bone remodeling during Radium therapy is correlated to overall survival and time to symptomatic skeletal event. Optimally these biomarkers can aid in monitoring therapy.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration resistant prostate cancer
* Planned to initiate Radium therapy
* Age > 18 years
* Able to understand study protocol and give informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic castration-resistant prostate cancer, who initiate therapy with Radium-223 at Rigshospitalet, Copenhagen, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Thrombocytopenia | Within 1 year from inclusion
  CTCAE grade 1-5
OS | within 1 year from inclusion
  Survival from first Radium-223
Bone markers | Within 12 months from inclusion
  Changes in bone metabolic markers during Radium-223

SECONDARY OUTCOMES:
Leucopenia | Within 1 year from inclusion
  CTCAE grade 1-5
Anemia | Within 1 year from inclusion
  CTCAE grade 3-5

CONTACTS AND LOCATIONS:
Overall Officials: Jann Ø Mortensen, DMSc, Study Director — Rigshospitalet, Department of Clinical Physiology, Nuclear Medicine & PET
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fosbol MO, Jorgensen NR, Petersen PM, Kjaer A, Mortensen J. Biomarkers of bone metabolism in [223Ra] RaCl2 therapy - association with extent of disease and prediction of overall survival. EJNMMI Res. 2024 Oct 3;14(1):90. doi: 10.1186/s13550-024-01155-w. PMID 39361218